CLINICAL TRIAL: NCT01738295
Title: Donepezil Effect on Visual Attention and Perceptual Training in Healthy Young Adults
Brief Title: Donepezil Effect on Visual Attention and Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Elvire Vaucher, Associate professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 12-084-CERES
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2015-08

CONDITIONS: Healthy
Keywords: acetylcholine; cholinergic system; visual perception; visual attention; multiple objects tracking; perceptual learning; vision training
MeSH Terms: interventions — Donepezil; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil (Active Comparator): Donepezil administration. In this group Donepezil (Aricept pill, 5 mg) will be orally administrated 3h before each experiment (1 week intervals)
  Interventions: Drug: Donepezil administration
- Lactose pill (Placebo Comparator): Placebo administration. In this group, placebo (lactose pill) will be orally administrated 3h before each experiments (1 week intervals)
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: Donepezil administration
  Other Names: Aricept, Pfizer
  Arms: Donepezil
Drug: Placebo administration
  Other Names: Lactose pill
  Arms: Lactose pill

SUMMARY:
The present proposal investigates the role of the cholinergic system (the neurotransmitter acetylcholine) in improving vision and visual attention. Vision results from a complex processing of particular stimuli of the visual field. Attention enhances and prolongs the neural representations of visual input in the visual cortex. It has recently been shown that attention in the visual cortex depends on cholinergic mechanisms. The action of acetylcholine in the visual cortex consists in enhancement of the responsiveness to thalamocortical inputs, depression of local neuronal connections or extrastriate feedback projections and induction of gamma synchronisation. The investigators hypothesize that these effects are associated with long-term changes in functional connectivity in the visual cortex, visual attention and visual learning (improvement of the visual capacities).

In the present proposal, the investigators will test whether the administration of donepezil (Aricept, 5mg), a drug that increases the level of acetylcholine in the brain, will enhances the perceptual-cognitive abilities of young adult subjects. Perceptual-cognitive performance will be assessed in a multiple object tracking (MOT) task in a 3D automatic virtual environment. MOT is a task where observers are asked to maintain attentional focus on a limited number of preselected subgroup of elements in a dynamic scene. Multifocal attentional mechanisms are necessary to process the information. The task will be tested five time at one week interval to test whether donepezil and training improved the task performance of the subject, i.e. lead to perceptual learning. This study could help establish an intervention procedure to improve visual performance of subjects that need it.

DETAILED DESCRIPTION:
Stages of a given perceptual-cognitive task (from Faubert and Sidebottom, Journal of Clinical Sport Psychology, 2012, 6, 85-102):

1. a predetermined number of spheres (typically eight) are presented in a 3D dimensional virtual volumetric cube space. The spheres are typically all identical.
2. a subset of spheres (typically four) is indexed via highlighting for a brief period of 1 s.
3. the spheres return to their original color and start moving within the restricted 3D virtual space. During this movement, the spheres can collide and consequently suddenly change direction, and they can cross over others, thus occluding their view.
4. the spheres stop moving after a predetermined time, and the observer has to identify the spheres that were initially indexed with halos. The subject is then given feedback on the response by having the spheres identified by revealing the appropriate indexed stimuli.

The main task starts at a given speed, and if all four spheres are not correctly identified, the next trial will be slower. If the four spheres are correctly identified, then the next trial will be faster. Trials are repeated like this following a staircase procedure, and ultimately, a speed threshold is established.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* 17 < body mass index < 25
* visual acuity 6/6
* visual stereoscopy > 50
* standard visual field

Exclusion Criteria:

* pregnancy or breast feeding
* use of any drug or St John's wort
* smoking
* asthma
* pulmonary obstruction
* cardiovascular impairment
* attention troubles
* ocular diseases
* epilepsy
* lactose intolerance
* absorption of grapefruit juice

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measure of the speed threshold, baseline | week 0
  The speed of the moving spheres is increased across trials until the subject is not able anymore to track and identify the indexed spheres (speed threshold). In this baseline task, the subject will not take Donepezil or placebo
Change from baseline of the speed threshold at 1 week | week 1
  The speed of the moving spheres is increased across trials. The maximal speed for which the subject is able to track and identify the indexed spheres is the speed threshold. At this time point, the effect of Donepezil (5 mg, single dose) or placebo administration on the perceptual-cognitive performance will be assessed.
Change from baseline of the speed threshold at 2 weeks | week 2
  The speed of the moving spheres is increased across trials. The maximal speed for which the subject is able to track and identify the indexed spheres is the speed threshold. At this time point, the effect of Donepezil (5 mg, single dose) or placebo administration on the perceptual-cognitive performance will be assessed.
Change from baseline of the speed threshold at 3 weeks | week 3
  The speed of the moving spheres is increased across trials. The maximal speed for which the subject is able to track and identify the indexed spheres is the speed threshold. At this time point, the effect of Donepezil (5 mg, single dose) or placebo administration on the perceptual-cognitive performance will be assessed.
Change from baseline of the speed threshold at 4 weeks | week 4
  The speed of the moving spheres is increased across trials. The maximal speed for which the subject is able to track and identify the indexed spheres is the speed threshold. At this time point, the effect of Donepezil (5 mg, single dose) or placebo administration on the perceptual-cognitive performance will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Elvire Vaucher, PhD, Study Director — Université de Montréal; Jocelyn Faubert, PhD, Study Director — Université de Montréal; Isabelle Legault, PhD, Principal Investigator — Université de Montréal; Mira Chamoun, MSc, Principal Investigator — Université de Montréal
Locations (1):
- School of optometry / Université de Montréal, Montreal, Quebec, Canada